CLINICAL TRIAL: NCT06356259
Title: A Randomised, Placebo-Controlled, Double-blind, Single and Multiple Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics Following Intravenous Administration of IRX-010 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics Following Intravenous Administration of IRX-010 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The highest multiple dose planned for this study was not well tolerated by most participants. There is no benefit to continue dosing of healthy participants.
Sponsor: ImmunoRx Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: IMMUNRX-01; 2023-503917-31 (EudraCT Number)
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IRX-010 Part A (SAD) (Experimental): A single dose of IRX-010 will be administered intravenously
  Interventions: Drug: IRX-010
- Placebo Part A (SAD) (Placebo Comparator): Placebo administered intravenously
  Interventions: Drug: Placebo
- IRX-010 Part B(MAD) (Experimental): Multiple doses of IRX-010 will be administered intravenously
  Interventions: Drug: IRX-010
- Placebo Part B(MAD) (Placebo Comparator): Placebo administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IRX-010 — Administered IV
  Arms: IRX-010 Part A (SAD); IRX-010 Part B(MAD)
Drug: Placebo — Administered IV
  Arms: Placebo Part A (SAD); Placebo Part B(MAD)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics with intravenous(IV) administration of IRX-010 in Healthy Participants.

DETAILED DESCRIPTION:
This is a single and multiple ascending dose, proof of concept study assessing the safe and tolerable dose of IRX-010 in healthy participants. Approximately 81 healthy participants will be enrolled in up to 9 cohorts. The study is conducted in two parts (part A and part B) with 6 single ascending dose (Part A - SAD) cohorts of 9 participants per cohort and 3 multiple ascending dose (Part B - MAD) cohorts of 9 participants per cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female participants who are healthy as determined by medical history and physical evaluation.
* Have clinical laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically. significant by the investigator at screening and enrolment.
* Have an estimated glomerular filtration rate ≥60 mL/minute/1.73 m2 at screening and enrolment.
* Have venous access sufficient to allow for blood sampling as per the protocol. Weight
* Have a body mass index of 18.0 to 32.0 kg/m2 inclusive, at screening.

Exclusion Criteria:

* Have a history or presence of clinically significant medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, haematological, renal, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicates a medical problem that would preclude study participation.
* Have history (within past 5 years) of, or presence of, uncontrolled asthma, significant rheumatological or autoimmune diseases, including but not limited to systemic lupus erythematosus, RA, Sjogren's Syndrome, or vasculitis; or hereditary angioedema, or common variable immune deficiency.
* Have had lymphoma, leukaemia, or any malignancy within the past 5 years.
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (if known) (whichever is longer) prior to dosing
* Have active or latent Tuberculosis (TB), based on a positive medical history, examination, chest x-rays (as per local TB screening guidelines), and/or TB test results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with Serious Adverse Events | Baseline upto Day 168
  Evaluation of Safety and Tolerability of IRX-010
Number of participants with Treatment-Emergent Adverse Events | Baseline upto Day 168
  Evaluation of Safety and Tolerability of IRX-010

SECONDARY OUTCOMES:
Pharmacokinetics(PK): Area under Curve(AUC) | Baseline upto Day 168
  PK: AUC of IRX-010
Pharmacokinetics(PK): Maximum Concentration (Cmax) | Baseline upto Day 168
  PK: Cmax of IRX-010
Pharmacokinetics(PK): Half-Life (t½) | Baseline upto Day 168
  PK: t½ of IRX-010

CONTACTS AND LOCATIONS:
Overall Officials: ImmunoRx Pharma,Inc, Study Director — ImmunoRx Pharma Inc.
Locations (1):
- ICON, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No